CLINICAL TRIAL: NCT02192723
Title: Effectiveness of 6 Antipsychotic Drugs in the Treatment of Acute Exacerbations of Chronic Inpatients With Schizophrenia: a Randomized Double-blind Study
Brief Title: A Randomized Double-blind Trial With 6 Antipsychotic Drugs for Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing HuiLongGuan Hospital (Other)
Responsible Party: Principal Investigator, Xiang Yang Zhang, Director, the Research Center, Beijing HuiLongGuan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Project863
Record Dates: First submitted 2014-07-15; First posted 2014-07-17 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Haloperidol; Perphenazine; Risperidone; Olanzapine; Quetiapine Fumarate; ziprasidone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Typical antipsychotic (Experimental): Haloperidol (6~20mg/day) and perphenazine (16~64mg/day) for 8 weeks.
  Interventions: Drug: Typical antipsychotic
- Risperidone (Active Comparator): Risperidone, 2~6mg/day, twice day, 8 weeks
  Interventions: Drug: Risperidone
- Olanzapine (Active Comparator): 5~20mg/day
  Interventions: Drug: Olanzapine
- Quetiapine (Active Comparator): 400~750mg/day
  Interventions: Drug: Quetiapine
- Aripiprazole (Active Comparator): Aripiprazole, 10~30mg/day, twice per day, 8 weeks
  Interventions: Device: Aripiprazole
- Ziprasidone (Active Comparator): Ziprasidone, 80~160mg/day, twice per day, 8 weeks
  Interventions: Drug: Ziprasidone

INTERVENTIONS:
Drug: Typical antipsychotic — Haloperidol (6~20mg/day) and perphenazine (16~64mg/day), twice per day, 8 weeks
  Other Names: Haldol and Trilafon
  Arms: Typical antipsychotic
Drug: Risperidone — 2~6mg/day, twice per day, 8 weeks
  Other Names: Risperdal
  Arms: Risperidone
Drug: Olanzapine — Olanzapine, 400~750mg/day, twice per day, 8 weeks
  Other Names: Zyprexa
  Arms: Olanzapine
Drug: Quetiapine — Quetiapine, 400～750mg/day, twice per day, 8 weeks
  Other Names: Seroquel
  Arms: Quetiapine
Device: Aripiprazole — Aripiprazole, 10～30mg/day, twice per day, 8 weeks
  Other Names: Abilify
  Arms: Aripiprazole
Drug: Ziprasidone — Ziprasidone 80~160mg/day, twice per day, 8 weeks
  Other Names: Geodon
  Arms: Ziprasidone

SUMMARY:
The purpose of this study is to compare the efficacy and side effects of 6 commonly used antipsychotic drugs in the treatment of schizophrenia in a Chinese population.

DETAILED DESCRIPTION:
The relative effectiveness of second-generation (atypical) antipsychotic drugs as compared with that of older agents has been incompletely addressed, though newer agents are currently used far more commonly. The investigators compared a first-generation antipsychotic, perphenazine or haloperidol, with several newer drugs in a double-blind study.

METHODS: A total of 550 patients with schizophrenia were recruited at 4 Chinese sites and randomly assigned to receive perphenazine (16 to 64 mg per day) or haloperidol(6 t0 20mg per day), olanzapine (5 to 20 mg per day), quetiapine (400 to 750 mg per day), aripiprazole (10 to 30 mg per day) or risperidone (2 to 6.0 mg per day) for up to 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients' diagnoses is based on the results of the Structured Clinical Interview for DSM (SCID) using the criteria of the fourth edition of the Diagnostic and Statistical Manual (DSM-IV), physical exams and routine chemistry, and hematology laboratory tests. Attending-level psychiatrists will use a Chinese translation of the SCID to interview patients and their family members, who are given freedom to ask additional questions if respondents do not understand the standard probes.
* Patients must meet the following criteria: (1) diagnosis of schizophrenia; (2) duration of illness more than 2 years; (3) between 25 and 60 years of age; and (5) have NOT received antipsychotic medication for at least 1 month;(6) acute exacerbations of chronic inpatients.
* A complete medical history, electroencephalograms and electrocardiogram are obtained, and a physical examination and laboratory tests are performed at study entrance. None of the study participants have abnormal findings on these tests.

Exclusion Criteria:

-

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 550 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | Baseline, 8 weeks

SECONDARY OUTCOMES:
Clinical Global Impression (CGI) | Baseline, 8 weeks
  The Clinical Global Impression rating scales are commonly used measures of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders

OTHER OUTCOMES:
Udvalg for Kliniske Undersogelser (UKU) Side Effect Rating Scale | Baseline, 8 weeks
  The UKU Side Effect Rating Scale is a comprehensive, clinician-rated scale, designed to assess the side effects in patients treated with psychotropic medications.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Ren Wang, MD, PhD, Study Director — Beijing HuiLongGuan Hospital
Locations (1):
- Beijing HuiLongGuan Hospital, Beijing, China